CLINICAL TRIAL: NCT06556836
Title: "Diagnostic Accuracy of Ultrasound Compared to Epidurography for Epidural Catheter Localization in Patients Undergoing Open Abdominal Surgery"
Brief Title: "Diagnostic Accuracy of Ultrasound Compared to Epidurography for Epidural Catheter Localization"
Status: Recruiting | Type: Observational
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Ana Garduño López, principal investigator (MSc and MD), Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Other Study IDs: ANE-4596-23-25-1
Record Dates: First submitted 2024-08-08; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Open Abdominal Surgery; Epidural Analgesia
Keywords: epidural catheter localization; epidural analgesia; open abdominal surgery; diagnostic accuracy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Doppler color and M-Mode ultrasound — A diagnostic test intervention using color Doppler and M-Mode ultrasound will be conducted to localize the catheter within the epidural space and compared with epidurography.
Device: Epidurography — An epidurography is an imaging procedure used to visualize the epidural space of the spine. The process involves inserting an epidural catheter, through which a contrast dye is injected. Fluoroscopy or X-rays are then used to capture real-time images of the contrast flow, helping to ensure the catheter's correct placement and to detect any localization anomalies. In this study, the epidurography will be performed in the radiology department by a radiologist and a pain management interventionist.

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of ultrasound for locating epidural catheters compared to the gold standard, epidurography. This study is focused on patients undergoing major open abdominal surgeries, who often experience moderate to severe pain during the first 24 to 48 hours after surgery.

The main questions it aims to answer are:

How does the accuracy of ultrasound for detecting epidural catheter placement compare to that of epidurography? Can ultrasound provide a reliable alternative to epidurography in surgical settings where epidurography is not feasible?

In this trial, participants will:

Undergo a standard epidural analgesia procedure for pain management during their surgery.

Have their epidural catheter placement checked using both ultrasound and epidurography.

Report their pain levels and any issues with pain control during the immediate postoperative period.

The study will assess whether ultrasound can effectively replace epidurography in confirming catheter placement, potentially offering a less invasive and more practical solution in routine surgical environments.

DETAILED DESCRIPTION:
Introduction

Major open abdominal surgeries often result in moderate to severe pain during the first 24-48 hours postoperatively. Epidural analgesia is effective in managing pain for open abdominal and thoracic surgeries during this immediate postoperative period and is considered the gold standard in accelerated rehabilitation protocols. The effectiveness of this pain relief method depends on the precise placement of the catheter in the epidural space. Since the procedure is performed blindly and relies on the anesthesiologist's skill, coupled with variations in anatomical structures, the failure rate of catheter placement ranges from 12% to 30%. Identifying catheter misplacement early in the postoperative period is challenging, as residual anesthetic effects may mask its ineffectiveness if the catheter is positioned outside the epidural space. This challenge can result in uncontrolled postoperative pain later on.

Given the inherent difficulties in catheter placement and the limitations of relying on indirect anatomical assessment and sensory cues, even experienced clinicians may find epidural catheter insertion challenging. Sensory testing and patient-reported pain scores, while useful, do not consistently offer objective confirmation of correct catheter placement. Therefore, more practical and objective methods are needed.

Ultrasound Techniques

Color Doppler ultrasound, which visualizes fluid dynamics and flow direction, and M-mode ultrasound, which provides grayscale images of movement, could offer valuable insights. When fluid is injected into a confined space like the epidural space, it is expected to create turbulence, which would appear as a burst of color on the Doppler image. This turbulence arises because the fluid encounters resistance as it moves through the narrow epidural space. Although studies have demonstrated the reliability of color Doppler ultrasound for visualizing fluid flow through a needle in the caudal space in both adults and children, this does not directly translate to assessing catheter placement in the lumbar epidural space. For example, case series by Riveros-Pérez et al. and Elsharkawy et al. reported that only 37% and 68% of epidural catheter tips were visible in the posterior complex using color Doppler, respectively. Studies have shown mixed results regarding their effectiveness, and their application to detecting catheter placement in the lumbar epidural space has yet to be fully established.

M-mode ultrasound, on the other hand, emits a single beam of ultrasound that traverses various structures, generating echoes that provide information on the mobility of different areas. This mode produces grayscale images where movement can be observed.

Epidurography

Epidurography, performed using radiographs, computed tomography, or fluoroscopy, remains the gold standard for verifying catheter placement when analgesia fails. This technique involves injecting an iodinated contrast agent through the catheter into the epidural space. The distribution of the contrast medium allows for visualization of the catheter's placement and verification of the correct vertebral level. Although epidurography provides definitive confirmation of catheter placement and helps mitigate patient dissatisfaction due to analgesic failure, it is less practical in the surgical setting due to the bulky equipment and the complexity of the procedure.

Safety of Contrast Medium in Epidurography Epidurography, which utilizes fluoroscopy, has been employed for several decades by interventional pain specialists. The incidence of adverse effects related to the contrast medium is extremely low, approximately 0.007%, due to the minimal volume of contrast required for the procedure.

Typically, epidurography involves the injection of 3 to 5 ml of iodinated contrast agent with a concentration of 240 mg/ml to verify accurate epidural placement. The rate of allergic reactions to iodinated contrast agents used in CT scans is estimated at around 0.6%, with severe reactions occurring in approximately 0.04% of cases. Most reactions are mild and can be managed or prevented with corticosteroids or small doses of adrenaline.

Radiation Exposure in Epidurography Radiation exposure is a critical consideration in ensuring patient safety. The effective radiation dose from fluoroscopic epidurography is approximately 1 mSv for a procedure lasting about 60 seconds. This dose is comparable to 10 days of natural background radiation exposure.

It is important to monitor both the duration of the procedure and the total radiation dose administered, which can be recorded by the imaging equipment.

Despite its extensive use and low-risk profile in interventional pain management, epidurography is not ideal for intraoperative settings, underscoring the need for more practical, real-time methods to ensure effective epidural analgesia.

Justification The literature has not yet established a systematic, objective method for evaluating the positioning of epidural catheters within the epidural space. Current research is exploring whether color Doppler and M-mode ultrasound could serve as reliable diagnostic tools for confirming correct catheter placement. Although alternative techniques like epidurography are available, they are less favored due to their requirement for bulky equipment and the exposure of patients to ionizing radiation. In contrast, ultrasound is a non-invasive and patient-safe option that is easy to learn and perform, offering high sensitivity and specificity.

Problem Statement In major abdominal surgeries performed under general anesthesia, combining epidural techniques with general anesthesia complicates the early evaluation of the catheter's sensory and analgesic blockade. This difficulty arises because residual pharmacological and anesthetic effects can alter the effectiveness of the neuraxial blockade analysis postoperatively. Delayed assessment of epidural analgesia can lead to significant issues in patient recovery, particularly due to the context-sensitive half-life of anesthetics and opioids, which may result in unmanaged pain hours later.

Hypothesis Research Question: What is the diagnostic accuracy of using ultrasound with Color Doppler Mode and M Mode for detecting the location of the epidural catheter in the epidural space compared to epidurography? Null Hypothesis (H0): The diagnostic accuracy of ultrasound using Color Doppler Mode and M Mode for detecting the location of the epidural catheter is less than 15% of the sensitivity of epidurography.

Alternative Hypothesis (H1): The diagnostic accuracy of ultrasound using Color Doppler Mode and M Mode for detecting the location of the epidural catheter is at least 15% of the sensitivity of epidurography.

Objectives Main Objective: Evaluate and compare the diagnostic accuracy of ultrasound using M-mode and color Doppler mode for locating the epidural catheter against epidurography.

Specific Objectives:

* Document and analyze demographic characteristics.
* Compare sonoanatomical distances and catheter positioning as determined by ultrasound in 2D Mode, M-mode, and color Doppler mode with those identified by epidurography.
* Determine and compare the diagnostic accuracy of ultrasound versus epidurography.
* Assess clinical and sensory block correlation with sensory tests and ultrasound findings.
* Measure analgesic efficacy using the verbal numerical scale (0-10) and the PAIN OUT international questionnaire (POD1).

Methods This study, approved by the Research and Ethics Committee of the Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, will be conducted at this tertiary hospital in Mexico City. This is a prospective, observational diagnostic test study aimed at evaluating and comparing the diagnostic accuracy of ultrasound (M-mode and color Doppler) versus epidurography for locating the epidural catheter. The study will involve the use of epidurography and ultrasound for each patient to assess diagnostic accuracy and is designed as a comparative study. Eligible patients will be provided with a detailed explanation of the study and will be required to sign written informed consent before participation.

Universe: Patients undergoing abdominal surgery requiring an epidural block for postoperative analgesia.

Observation Units: Each patient scheduled for abdominal surgery requiring an epidural block.

Sampling Method: Recruitment based on the need for an epidural block for postoperative analgesia.

Data Collection

Ultrasound and Epidurography While the patient remains in the post-anesthesia care unit (PACU), an initial ultrasound assessment will be conducted by a trained anesthesiologist from the acute pain service. This scan will last between 15 and 30 minutes, and the observer will record the findings using a Google Form.

Upon discharge from the PACU, an epidurography will be performed in the radiology department, where a radiologist and an interventional pain physician will be available to conduct and interpret the results of the epidurography.

Following the epidurography, another ultrasound scan will be conducted by a second trained anesthesiologist from the acute pain service to evaluate interobserver variability.

Sensitivity Assessment Within the first 6 hours post-procedure, the acute pain management team will evaluate the sensitivity of the dermatomes corresponding to the surgical wound on the abdominal wall at the bedside.

Two methods will be employed for this sensitivity assessment: pinprick (using a blunt needle for point stimulation) and cold pressure (applying a cotton swab with alcohol).

These assessments will be conducted symmetrically, beginning with the T5 dermatome and progressing in a caudal direction along the abdominal wall to define the region of reduced sensitivity.

Assessment of Pain at Rest and Dynamic Pain To evaluate pain characteristics and patient satisfaction, the international PAIN OUT questionnaire will be administered 24 hours after the procedure. This questionnaire will help in assessing both pain at rest and dynamic pain levels experienced by the patient.

Scanning Protocol: A scanning protocol, developed and refined since January 2023, will be followed for the study. This protocol outlines the methodology for performing the ultrasound scans in our Institute.

Ultrasound with Color Doppler Mode and M-Mode: A Sonosite Nanomax ultrasound device equipped with a 2-5 MHz curved probe will be used. This device includes both Color Doppler mode and M-mode capabilities, enabling real-time visualization of the epidural catheter's position and assessment of flow distribution within the epidural space.

Epidurography Equipment in the Radiology Area: Fluoroscopy equipment will be employed to perform epidurography. This involves injecting a contrast agent (Iopamidol, 3-5 milliliters) into the epidural space to obtain images that assess the catheter's positioning.

Data Recording Equipment: Data will be systematically recorded using a Google Form. This system will collect and store all relevant information obtained during the study, including ultrasound data, epidurography results, and other pertinent details necessary for subsequent analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Provided informed consent
* Scheduled for major open abdominal surgery that necessitates epidural analgesia
* Capable of completing the PAIN OUT questionnaire

Exclusion Criteria:

* Contraindications to epidural analgesia
* Communication or cognitive impairments that prevent understanding or completing the questionnaire
* Neurological disorders that affect sensory or motor function
* Critical illness or unstable medical conditions
* Use of anticoagulants
* Advanced liver cirrhosis
* Certain specific surgical procedures where epidural analgesia is contraindicated or not applicable
* Allergy to contrast agent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both sexes, aged 18 and over, who provide informed consent, scheduled for major open abdominal surgery requiring epidural analgesia at the Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, will be approached for participation. Inclusion and exclusion criteria will be applied to identify eligible participants. Those who meet the criteria and provide informed consent will be enrolled in the study. The sample size will be adjusted to ensure that 50 patients are recruited.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of ultrasound color Doppler compared to epidurography for localizing the catheter in the epidural space. | 15 minutes
  Ultrasound Doppler Mode: To assess whether the color mosaic between the posterior and anterior complexes is observed when saline solution is administered through the catheter, indicating correct placement within the epidural space.
  Epidurography: Performed by an interventional pain specialist and a radiologist, it will confirm whether the catheter is correctly positioned inside or outside the epidural space.
  Diagnostic Accuracy of Ultrasound: Evaluated by comparing the findings from Doppler mode and M-mode (color mosaic and granular pattern) with the results of epidurography (inside or outside the epidural space).
Diagnostic accuracy of ultrasound Mode M compared to epidurography for localizing the catheter in the epidural space. | 15 minutes
  Ultrasound M-Mode: To detect a granular or undulating pattern when intermittent boluses of saline solution are administered through the epidural catheter, which indicates correct placement within the epidural space.

SECONDARY OUTCOMES:
Pain Relief Effectiveness | 10 to 15 minutes
  At 24 hours postoperatively, patients will complete an internationally validated and standardized questionnaire to assess static and dynamic pain intensity. This questionnaire includes 13 questions that evaluate various aspects of the patient's experience. These aspects include static and dynamic pain, adverse effects, anxiety, overall pain, perception of care, satisfaction, and history of chronic pain.
Sensory Assessment Level of Abdominal Wall: | 5 minutes
  Assessment Technique: Utilize a standardized method, such as a pinprick test, cotton swab, or temperature sensation test, to evaluate sensory responses across different regions of the abdominal wall

CONTACTS AND LOCATIONS:
Overall Officials: ANA LILIA GARDUÑO-LOPEZ, M.Sc, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; GUSTAVO LUGO-GOYTIA, D.Sc, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Tlalpan, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Elsharkawy H, Sonny A, Govindarajan SR, Chan V. Use of colour Doppler and M-mode ultrasonography to confirm the location of an epidural catheter - a retrospective case series. Can J Anaesth. 2017 May;64(5):489-496. doi: 10.1007/s12630-017-0819-y. Epub 2017 Jan 10. PMID 28074426
- [Result] Riveros-Perez E, Albo C, Jimenez E, Cheriyan T, Rocuts A. Color your epidural: color flow Doppler to confirm labor epidural needle position. Minerva Anestesiol. 2019 Apr;85(4):376-383. doi: 10.23736/S0375-9393.18.13175-0. Epub 2018 Nov 22. PMID 30482003
- [Result] van den Bosch OFC, Gleicher Y, Arzola C, Siddiqui N, Downey K, Carvalho JCA. Color flow Doppler in spinal ultrasound: a novel technique for assessment of catheter position in labor epidurals. Reg Anesth Pain Med. 2022 Dec;47(12):775-779. doi: 10.1136/rapm-2022-103948. Epub 2022 Sep 7. PMID 36215115
- [Result] Coleman JR, Hartmann P, Kona M, Thiele RA, Salajegheh R, Hanson NA. Use of epidurography in the perioperative and acute pain setting. Reg Anesth Pain Med. 2022 Jul;47(7):445-448. doi: 10.1136/rapm-2021-103274. Epub 2022 Apr 20. PMID 35443993
- [Result] Hermanides J, Hollmann MW, Stevens MF, Lirk P. Failed epidural: causes and management. Br J Anaesth. 2012 Aug;109(2):144-54. doi: 10.1093/bja/aes214. Epub 2012 Jun 26. PMID 22735301
- [Result] Weiss R, Popping DM. Is epidural analgesia still a viable option for enhanced recovery after abdominal surgery. Curr Opin Anaesthesiol. 2018 Oct;31(5):622-629. doi: 10.1097/ACO.0000000000000640. PMID 29994937
- [Result] Garduno-Lopez AL, Acosta Nava VM, Castro Garces L, Rascon-Martinez DM, Cuellar-Guzman LF, Flores-Villanueva ME, Villegas-Sotelo E, Carrillo-Torres O, Vilchis-Samano H, Calderon-Vidal M, Islas-Lagunas G, Richard Chapman C, Komann M, Meissner W, Baumbach P, Zaslansky R. Towards Better Perioperative Pain Management in Mexico: A Study in a Network of Hospitals Using Quality Improvement Methods from PAIN OUT. J Pain Res. 2021 Feb 15;14:415-430. doi: 10.2147/JPR.S282850. eCollection 2021. PMID 33623424
- [Result] PAIN OUT Research Group Jena; Chinese PAIN OUT network; Dutch PAIN OUT network; Mexican PAIN OUT network; Serbian PAIN OUT network; Spanish PAIN OUT network; French PAIN OUT network; Italian PAIN OUT network; Swiss PAIN OUT network; Irish PAIN OUT network; Belgian PAIN OUT network; Zaslansky R. Status quo of pain-related patient-reported outcomes and perioperative pain management in 10,415 patients from 10 countries: Analysis of registry data. Eur J Pain. 2022 Nov;26(10):2120-2140. doi: 10.1002/ejp.2024. Epub 2022 Sep 26. PMID 35996995
- See also: Garduño-López AL,et al.Optimization of epidural analgesia: proposed protocol for evaluation with Doppler Ultrasound and M Mode for precise catheter localization.Rev Mex Anestesiol. 2024; 47 (4): 236-242. https://dx.doi.org/10.35366/116229 — https://dx.doi.org/10.35366/116229